CLINICAL TRIAL: NCT06775769
Title: Endometrioma Sclerotherapy and Ovarian Preservation: a Randomised Control Trial of Laparoscopic Sclerotherapy vs Traditional Excision of Endometrioma
Brief Title: Endometrioma Sclerotherapy and Ovarian Preservation
Acronym: ENDOSAVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24/LO/0825
Record Dates: First submitted 2024-12-12; First posted 2025-01-15 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Endometrioma
Keywords: Endometrioma; Endometriosis; Sclerotherapy
MeSH Terms: conditions — Endometriosis | interventions — Sclerotherapy

STUDY DESIGN:
Intervention Model Description: Randomised control trial
Who Masked: Participant
Masking Description: Ultra-sonographer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical Management of Endometrioma (Other): Routine Care
  Interventions: Procedure: Routine Care
- Laparoscopic Sclerotherapy (Experimental): Laparoscopic ethanol sclerotherapy of endometrioma
  Interventions: Procedure: Sclerotherapy

INTERVENTIONS:
Procedure: Sclerotherapy — Laparoscopic ethanol sclerotherapy of endometrioma
  Arms: Laparoscopic Sclerotherapy
Procedure: Routine Care — Routine surgical management of endometrioma
  Arms: Surgical Management of Endometrioma

SUMMARY:
A randomised controlled trial assessing ovarian reserve after laparoscopic ethanol sclerotherapy of ovarian endometrioma compared to standard treatment of surgical excision of endometrioma.

Secondary outcomes will include endometrioma recurrence, symptomatology and inflammatory environment.

DETAILED DESCRIPTION:
Participants with endometrioma(ta), identified on imaging, who are opting for surgical management of endometriosis will be randomly allocated to laparoscopic ethanol sclerotherapy of endometrioma or laparoscopic surgical excision of endometrioma(ta). Any concurrent endometriosis identified at surgery will be excised as per routine care.

Ovarian reserve will be assessed by serum anti-Mullarian hormone (AMH) and antral follicle count (AFC), recurrence will me assessed by transvaginal ultrasound, symptomatology will be assessed by EHP-30 questionnaires and changes in inflammation assessed in serum and endometrial biopsy.

Each participant will be followed up for a total of 24 months from surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female (XX genotype, assigned female at birth)
* Age 18-40
* Finding of suspected uni- or bi-lateral ovarian endometrioma(ta) of ≥ 2cm on TVUSS and/or pelvic MRI scan (TVUSS, a uni- or multi-locular ovarian cystic lesion with low level echoes and diffuse homogeneous ground glass appearance; MRI any of, ovarian lesion hyperintense T1 without loss of signal on T1 fat-suppressed images, hypointense T2 exhibiting shading sign and/or T2 dark spot sign, variable restricted diffusion on DWI)
* Appropriate to be listed for laparoscopic excision of endometrioma (Endometrioma ≥2cm, pain symptoms attributable to endometriosis where medical management is unsuccessful or unacceptable to the patient, to facilitate ART)

Exclusion Criteria:

* Postmenopausal status
* Suspicion of malignancy
* Unable to undergo TVUSS
* Declines to take part in the study
* Unable to understand verbal or written information in English
* Lack of capacity to consent at the point of recruitment
* Known safeguarding issues

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Ovarian Reserve | 24 months
  To determine the statistical difference in ovarian reserve pre- and post- treatment (as measured by serum AMH at 3, 6, 12 and 24 months and antral follicle count at 6, 12 and 24 months) in participants randomised to receive laparoscopic ethanol sclerotherapy or laparoscopic excision of endometrioma

SECONDARY OUTCOMES:
Endometrioma recurrence | 24 monhts
  To determine if laparoscopic ethanol sclerotherapy for ovarian endometrioma alters recurrence of ovarian endometrioma (as measured by TVUSS at 6, 12 and 24 months) as compared to laparoscopic excision of endometrioma
Symptomatology | 24 monhts
  To determine if laparoscopic ethanol sclerotherapy for ovarian endometrioma affects symptomatology (as recorded by EHP-30) as compared to laparoscopic excision of endometrioma at 3, 6, 12 and 24 months
Inflammation | 24 monhts
  To determine if laparoscopic ethanol sclerotherapy for ovarian endometrioma alters the inflammatory environment (as measured in blood at 3, 6, 12 and 24 months, and endometrial biopsy at 6 months) as compared to laparoscopic excision of endometrioma

CONTACTS AND LOCATIONS:
Locations (1):
- Chelsea and Westminster NHS Foundation Trust, London, United Kingdom